CLINICAL TRIAL: NCT02061358
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single-Ascending Dose Study to Determine the Safety, Tolerability and Pharmacokinetics of UV-4B Solution Administered Orally in Healthy Subjects
Brief Title: Study to Determine the Safety, Tolerability and Pharmacokinetics of UV-4B Solution Administered Orally in Healthy Subjects
Acronym: UV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Quintiles, Inc. (Industry); Unither Virology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMID 13-0001; KQA71264; UV-DEN-0001
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Viral Infection
Keywords: Dengue; Arbovirus Infections; Flaviviridae Infections; Flavivirus Infections; Hemorrhagic Fevers, Viral; RNA Virus Infections; Virus Diseases; Pharmaceutical Solutions; Pharmacologic Actions; Therapeutic Uses
MeSH Terms: conditions — Virus Diseases; Dengue; Arbovirus Infections; Flaviviridae Infections; Flavivirus Infections; Hemorrhagic Fevers, Viral; RNA Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1 - 3 mg UV-4B (Experimental): Subjects receiving UV-4B 3 mg oral solution or placebo
  Interventions: Drug: UV-4B 3 mg; Drug: Placebo
- Cohort 2 - 10 mg UV-4B (Experimental): Subjects receiving UV-4B 10 mg oral solution or placebo
  Interventions: Drug: UV-4B 10 mg; Drug: Placebo
- Cohort 3- 30 mg UV-4B (Experimental): Subjects receiving UV-4B 30 mg oral solution or placebo
  Interventions: Drug: UV-4B 30 mg; Drug: Placebo
- Cohort 4 - 90 mg UV-4B (Experimental): Subjects receiving UV-4B 90 mg oral solution or placebo
  Interventions: Drug: UV-4B 90 mg; Drug: Placebo
- Cohort 5 - 180 mg UV-4B (Experimental): Subjects receiving UV-4B 180 mg oral solution or placebo
  Interventions: Drug: UV-4B 180 mg; Drug: Placebo
- Cohort 6 - 360 mg UV-4B (Experimental): Subjects receiving UV-4B 360 mg oral solution or placebo
  Interventions: Drug: UV-4B 360 mg; Drug: Placebo
- Cohort 7 - 720 mg UV-4B (Experimental): Subjects receiving UV-4B 720 mg oral solution or placebo
  Interventions: Drug: UV-4B 720 mg; Drug: Placebo
- Cohort 8 - 1000 mg UV-4B (Experimental): Subjects receiving UV-4B 1000 mg oral solution or placebo
  Interventions: Drug: UV-4B 1000 mg; Drug: Placebo

INTERVENTIONS:
Drug: UV-4B 3 mg — Oral solution, single dose
  Arms: Cohort 1 - 3 mg UV-4B
Drug: UV-4B 10 mg — Oral solution, single dose
  Arms: Cohort 2 - 10 mg UV-4B
Drug: UV-4B 30 mg — Oral solution, single dose
  Arms: Cohort 3- 30 mg UV-4B
Drug: UV-4B 90 mg — Oral solution, single dose
  Arms: Cohort 4 - 90 mg UV-4B
Drug: UV-4B 180 mg — Oral solution, single dose
  Arms: Cohort 5 - 180 mg UV-4B
Drug: UV-4B 360 mg — Oral solution, single dose
  Arms: Cohort 6 - 360 mg UV-4B
Drug: UV-4B 720 mg — Oral solution, single dose
  Arms: Cohort 7 - 720 mg UV-4B
Drug: UV-4B 1000 mg — Oral solution, single dose
  Arms: Cohort 8 - 1000 mg UV-4B
Drug: Placebo — Oral solution, single dose

SUMMARY:
The objective is to evaluate the safety and tolerability of a single-ascending oral dose of UV-4B in healthy subjects and to determine pharmacokinetic parameters describing absorption and elimination following a single dose of UV-4B in healthy subjects.

DETAILED DESCRIPTION:
The causative agent of dengue fever is Dengue Virus (DENV), a member of the flavivirus genus. There are four DENV serotypes. Infection with one serotype results in lifelong immunity against that serotype, but only limited short-term cross-protection from infection with the other serotypes. Immunity to one serotype has a downside as subsequent infections by other serotypes increase the risk of developing more severe forms of dengue, which includes the most lethal form of the disease, dengue hemorrhagic fever. Traditional epidemiologic and serologic-based estimates suggest a range of 50 to 100 million DENV infections per year distributed over 100 countries. Recent cartographic-based modeling studies suggest that up to 390 million of dengue infections per year, of which 96 million are associated with clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Women: non-pregnant, non-lactating; if of childbearing potential, on specified contraception measures during the study period
* Men: using barrier contraception measures during the study period

Exclusion Criteria:

* Health conditions
* Taking prescription and non-prescription drugs (exceptions: acetaminophen, vitamins, hormonal birth control)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Murtaugh, Dr, Principal Investigator — Senior Medical Research Director, Quintiles
Locations (1):
- Quintiles, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Callahan M, Treston AM, Lin G, Smith M, Kaufman B, Khaliq M, Evans DeWald L, Spurgers K, Warfield KL, Lowe P, Duchars M, Sampath A, Ramstedt U. Randomized single oral dose phase 1 study of safety, tolerability, and pharmacokinetics of Iminosugar UV-4 Hydrochloride (UV-4B) in healthy subjects. PLoS Negl Trop Dis. 2022 Aug 8;16(8):e0010636. doi: 10.1371/journal.pntd.0010636. eCollection 2022 Aug. PMID 35939501
- See also: Information on dengue fever — http://www.niaid.nih.gov/topics/denguefever/Pages/default.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single center study performed in the United States. The study was completed with a total of 64 patients enrolled.
Pre-assignment Details: Each cohort was assigned 6 subjects who received the cohort's prescribed dose of UV-4B, along with 2 subjects in each cohort assigned to receive placebo.
Groups:
- 3 mg UV-4B: UV-4B 3 mg oral, single dose
- 10 mg UV-4B: UV-4B 10 mg oral, single dose
- 30 mg UV-4B: UV-4B 30 mg oral, single dose
- 90 mg UV-4B: UV-4B 90 mg oral, single dose
- 180 mg UV-4B: UV-4B 180 mg oral, single dose
- 360 mg UV-4B: UV-4B 360 mg oral, single dose
- 720 mg UV-4B: UV-4B 720 mg oral, single dose
- 1000 mg UV-4B: UV-4B 1000 mg oral, single dose
- Placebo: Placebo oral, single dose
Period: Overall Study
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number of randomized subjects in each cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5) | 27 (8) | 27 (4) | 28 (9) | 28 (9) | 29 (9) | 25 (9) | 27 (8) | 28 (8) | 27 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 1 | 1 | 3 | 1 | 3 | 17
  Male | 3 | 4 | 4 | 5 | 5 | 5 | 3 | 5 | 13 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 9
  Not Hispanic or Latino | 5 | 5 | 6 | 5 | 3 | 6 | 6 | 5 | 14 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 2 | 1 | 2 | 2 | 0 | 2 | 12
  White | 6 | 3 | 5 | 4 | 5 | 4 | 4 | 6 | 14 | 51
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 173.4 (11.1) | 171.8 (12.3) | 175.0 (11.3) | 175.2 (3.8) | 176.2 (9.9) | 174.8 (8.9) | 172.6 (8.2) | 173.5 (3.2) | 174.9 (8.1) | 174.25 (8.39)
Weight [Mean (Standard Deviation); unit: kg] | 82.9 (12.1) | 79.6 (13.8) | 80.8 (9.7) | 75.9 (8.3) | 84.0 (8.5) | 80.1 (10.5) | 74.1 (11) | 75.0 (5.5) | 76.2 (11.5) | 78.36 (10.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.44 (1.28) | 26.88 (2.6) | 26.44 (2.36) | 24.76 (2.71) | 27.05 (1.84) | 26.13 (2.07) | 24.86 (2.93) | 24.93 (1.6) | 24.89 (2.82) | 25.77 (2.47)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Treatment-emergent Adverse Event (TEAEs) by Treatment Group
Description: TEAEs are those AEs occurring only after administration of investigational product
Time Frame: From time of the first dose administration through Day 9 ± 1
Population: Safety Population: all subjects who received any investigational product, UV-4B or placebo
Measure: Number; unit: Subjects with at least 1 TEAE
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Subjects with at least 1 TEAE | 5 | 6 | 5 | 5 | 6 | 5 | 6 | 5 | 12

2. Primary Outcome: Subjects With Serious Adverse Event (SAEs) by Treatment Group
Description: Subjects with AEs considered serious by the investigator
Time Frame: From time of the first dose administration through Day 9 ± 1
Population: Safety Population: all subjects who received any investigational product, UV-4B or placebo
Measure: Number; unit: Subjects with at least 1 SAE
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Subjects with at least 1 SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Vital Sign Values of Toxicity Grade 1 or Higher Postdose by Treatment Group (Safety Population)
Description: Number of subjects in a treatment group, who had a vital sign value of toxicity Grade 1 or higher: supine and standing systolic blood pressure (BP), supine and standing diastolic BP, supine and standing pulse rate, respiratory rate, and temperature
Time Frame: From time of the first dose administration through Day 9 ± 1
Population: Safety Population: all subjects who received any investigational product, UV-4B or placebo
Measure: Number; unit: Participants
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Participants
  Subjects with any Grade 1 or higher | 6 | 6 | 5 | 5 | 6 | 5 | 6 | 6 | 12
  Supine systolic BP ≤ 89 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Supine systolic BP ≥ 141 mmHg | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Standing systolic BP ≤ 89 mmHg | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Standing systolic BP ≥ 141 mmHg | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 1
  Supine diastolic BP ≥ 91 mmHg | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Standing diastolic BP ≥ 91 mmHg | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 1 | 3
  Supine pulse ≤ 50 bpm, baseline ≤ 60 bpm | 0 | 3 | 1 | 2 | 1 | 1 | 1 | 3 | 4
  Supine pulse ≤ 54 bpm, baseline > 60 bpm | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1
  Supine pulse ≥ 101 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Standing pulse ≤ 50 bpm, baseline ≤ 60 bpm) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing pulse ≤ 54 bpm, baseline > 60 bpm | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Standing pulse ≥ 101 bpm | 6 | 6 | 2 | 3 | 5 | 4 | 6 | 4 | 9
  Respiratory rate ≥ 17 breaths/min | 3 | 4 | 1 | 2 | 3 | 1 | 3 | 2 | 5
  Temperature ≥ 100.4 ⁰F (38.0 ⁰C) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Subjects With Electrocardiogram Outlier Values Postdose by Treatment Group
Description: Number of subjects in a treatment group with outlier ECG findings: QTcF (Fridericia's), PR, and QRS intervals
Time Frame: From time of the first dose administration through Day 9 ± 1
Population: Safety Population: all subjects who received any investigational product, UV-4B or placebo
Measure: Number; unit: participants
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
participants
  Subjects with an outlier value | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF > 450 ms (males) or > 470 ms (females) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF > 500 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF increase from baseline > 30 ms or ≤ 60 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF increase from baseline > 220 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR > 220 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS > 120 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Clinical Laboratory Test Results of Toxicity Grade 1 or Higher at Day 9 by Treatment Group
Description: Number of subjects with Grade 1 toxicity or higher for hematology, coagulation, chemistry and urinalysis analytes. ULN=upper limit of normal; WBC=white blood cell count.
Time Frame: Day 9 ± 1
Population: Safety Population: all subjects who received any investigational product, UV-4B or placebo
Measure: Number; unit: Participants
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Participants
  Hemoglobin ≤ 11.5 (♀), 13.5 (♂) g/dL or any ↓ | 3 | 5 | 5 | 4 | 4 | 3 | 3 | 3 | 14
  WBC ≥ 10,800 or ≤ 3,500 cell/mm^3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Neutrophils ≤ 2,000 cell/mm^3 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2
  Lymphocytes ≤ 1,000 cell/mm^3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils ≥ 650 cell/mm^3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Prothrombin time ≥ 1 * ULN | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time ≥ 1 * ULN | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Alkaline phosphatase ≥ 2 * ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase ≥ 1.1 * ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Aspartate aminotransferase ≥ 1.1 * ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bilirubin ≥ 1.1 * ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium ≤ 8.8 or ≥ 10.6 mg/dL | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 0
  Magnesium ≤ 1.7 mg/dL | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphorous ≤ 2.5 mg/dL | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Potassium ≤ 3.5 or ≥ 5.3 mEq/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Sodium ≤ 134 or ≥ 148 mEq/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin ≤ 3.3 g/dL | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total protein ≤ 5.9 g/dL | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Blood urea nitrogen ≥ 21 mg/dL | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine ≥ 1.5 mg/dL | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose ≤ 69 or ≥100 (fasting)/111 (random) mg/dL | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Creatine phosphokinase ≥ 2 * ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Amylase ≥ 1.5 * ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase ≥ 1.5 * ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose trace or more | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine protein trace or more | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Urine red blood cell count ≥ 1 rbc/hpf | 2 | 4 | 3 | 3 | 1 | 2 | 5 | 3 | 10

6. Secondary Outcome: Cmax by Treatment Group: UV-4
Description: Cmax is the maximum plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: Blood samples were collected at predose (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 18, 24, 36, and 48 hours postdose (1 hour window for predose)
Population: The pharmacokinetic (PK) population consisted of all subjects who received active investigational product, UV-4B, and had at least 1 measured concentration at a scheduled PK time after start of dosing for UV-4B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 22.1 (15.4) | 82.6 (24.2) | 289 (17.5) | 900 (35.3) | 2060 (33.6) | 4490 (20.0) | 9760 (20.0) | 13000 (15.6)

7. Secondary Outcome: Tmax by Treatment Group: UV-4
Description: Tmax is the time of maximum concentration observed directly from the observed concentration versus time data.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 0.50 [0.50 to 1.0] | 1.00 [0.50 to 1.50] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.52] | 0.75 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 1.00 [0.50 to 1.50]

8. Secondary Outcome: AUC(0-last) by Treatment Group: UV-4
Description: AUC(0-last) is the area under the concentration-time curve from time zero (pre-dose) to time of last quantifiable concentration, calculated by linear up/log down trapezoidal summation.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h/mL
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng * h/mL | 82.1 (18.8) | 406 (24.7) | 1230 (10.9) | 3640 (12.7) | 7050 (8.3) | 13600 (14.6) | 32700 (10.9) | 42700 (13.2)

9. Secondary Outcome: AUC(0-inf) by Treatment Group: UV-4
Description: AUC(0-inf) is the area under the concentration-time curve in the sample from pre-dose extrapolated to infinite time, calculated by linear up/log down trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration divided by the apparent terminal rate constant: AUC(0-last) - C(last)/λ(z).
Time Frame: as for outcome 6
Population: The pharmacokinetic (PK) population consisted of all subjects who received active investigational product, UV-4B, and had at least 1 measured concentration at a scheduled PK time after start of dosing for UV-4B. Subjects in this population were used for all PK summaries.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h/mL
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng * h/mL | 94.6 (16.3) | 420 (24.2) | 1260 (10.2) | 3700 (13.3) | 7090 (8.2) | 13700 (14.6) | 32800 (10.9) | 42800 (13.3)

10. Secondary Outcome: CL/F by Treatment Group: UV-4
Description: CL/F is the apparent systematic clearance, calculated as dose (free-base equivalent) divided by AUC(0-inf).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h | 31.7 (16.3) | 23.8 (24.1) | 23.9 (10.5) | 24.3 (13.5) | 25.4 (8.2) | 26.3 (14.7) | 22.0 (11.0) | 23.4 (13.3)

11. Secondary Outcome: Vz/F by Treatment Group: UV-4
Description: Vz/F is the apparent volume of distribution of UV-4 based on the terminal phase, calculated as dose (free-base equivalent) divided by [λ(z) × AUC(0-inf)].
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L | 470 (32.8) | 409 (30.6) | 344 (16.7) | 358 (21.5) | 317 (17.2) | 308 (11.9) | 259 (10.3) | 290 (27.3)

12. Secondary Outcome: t(1/2) by Treatment Group: UV-4
Description: t(1/2) is the apparent terminal half-life, determined as ln(2)/λ(z).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 9.11 [7.75 to 16.3] | 11.6 [10.6 to 13.7] | 9.98 [8.75 to 10.8] | 9.56 [8.52 to 16.0] | 8.52 [7.65 to 10.3] | 8.14 [7.06 to 9.08] | 8.03 [7.66 to 9.23] | 7.95 [6.60 to 13.4]

13. Secondary Outcome: Interval and Cumulative Amount (mg) of UV-4 Excreted in Urine, Ae, by Treatment Group
Description: Ae is the by-interval and cumulative amounts of UV-4 drug excreted in urine. Intervals were 0 to 6, 6 to 12, 12 to 24, and 24 to 48 hours postdose. Ae by-interval amounts were calculated as the product of urine volume and urine concentration. Ae(0-last) is the cumulative amount of UV-4 drug excreted in urine over the entire collection period, 48 hours. Cumulative amounts were calculated as the summation of the amounts excreted in collection intervals.
Time Frame: Pooled urine samples were collected at predose (-12 to 0 hour), and from 0 to 6, 6 to 12, 12 to 24, and 24 to 48 hours postdose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg
  Ae(0-6) | 0.607 (0.145) | 2.67 (0.386) | 10.6 (1.18) | 38.1 (3.83) | 77.5 (3.49) | 159 (24.3) | 301 (36.3) | 428 (64.5)
  Ae(6-12) | 0.215 (0.0496) | 0.859 (0.112) | 2.45 (0.145) | 6.05 (2.55) | 12.1 (1.48) | 19.1 (7.00) | 42.5 (6.00) | 53.7 (15.2)
  Ae(12-24) | 0.202 (0.0543) | 0.608 (0.0888) | 1.61 (0.363) | 3.89 (0.799) | 6.06 (2.40) | 7.09 (1.90) | 11.7 (1.60) | 16.4 (5.32)
  Ae(24-48) | 0.170 (0.0416) | 0.503 (0.0655) | 0.887 (0.200) | 1.61 (0.474) | 2.43 (1.03) | 2.83 (0.672) | 4.09 (1.24) | 5.21 (1.41)
  Ae(0-12) | 0.822 (0.177) | 3.53 (0.428) | 13.0 (1.31) | 44.1 (3.83) | 89.6 (3.76) | 178 (18.7) | 355 (34.6) | 498 (65.6)
  Ae(0-24) | 1.02 (0.197) | 4.13 (0.515) | 14.6 (1.13) | 48.0 (3.75) | 95.7 (4.26) | 185 (17.9) | 355 (34.6) | 498 (65.6)
  Ae(0-last) | 1.19 (0.200) | 4.64 (0.463) | 15.5 (0.982) | 49.6 (3.58) | 97.9 (4.86) | 188 (17.3) | 360 (34.7) | 504 (66.1)

14. Secondary Outcome: Interval and Cumulative Percent of UV-4 Excreted in Urine, fe, by Treatment Group
Description: fe is the by-interval percentage of UV-4 drug excreted in urine. Intervals were 0 to 6, 6 to 12, 12 to 24, and 24 to 48 hours postdose. fe = Ae/(UV-4B dose x 100). fe(0-12), fe(0-24) and fe(0-last) are the cumulative percentages of UV-4 drug excreted in urine over 24 hours and the entire collection period, respectively.
Time Frame: as for outcome 13
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of dose
  fe(0-6) | 20.2 (4.81) | 26.7 (3.86) | 35.3 (3.84) | 42.2 (4.26) | 43.0 (1.96) | 44.2 (6.69) | 41.8 (5.04) | 42.8 (6.45)
  fe(6-12) | 7.17 (1.65) | 8.59 (1.12) | 8.16 (0.480) | 6.72 (2.83) | 6.74 (0.820) | 5.32 (1.94) | 5.90 (0.833) | 5.37 (1.52)
  fe(12-24) | 6.71 (1.82) | 6.08 (0.888) | 5.36 (1.21) | 4.32 (0.886) | 3.37 (1.34) | 1.97 (0.532) | 1.63 (0.221) | 1.64 (0.532)
  fe(24-48) | 5.66 (1.39) | 5.03 (0.655) | 2.96 (0.664) | 1.79 (0.528) | 1.35 (0.572) | 0.787 (0.186) | 0.569 (0.172) | 0.521 (0.141)
  fe(0-12) | 27.4 (5.93) | 35.3 (4.28) | 43.4 (4.28) | 49.0 (4.28) | 49.8 (2.08) | 49.5 (5.18) | 47.7 (4.86) | 48.2 (6.66)
  fe(0-24) | 34.1 (6.57) | 41.3 (5.15) | 48.8 (3.72) | 53.3 (4.14) | 53.1 (2.37) | 51.5 (4.97) | 49.4 (4.81) | 49.8 (6.56)
  fe(0-last) | 39.8 (6.66) | 46.4 (4.63) | 51.7 (3.27) | 55.1 (3.98) | 54.5 (2.76) | 52.3 (4.82) | 49.9 (4.84) | 50.4 (6.61)

15. Secondary Outcome: CLr by Treatment Group: UV-4
Description: CLr is the renal clearance, calculated at Ae(0-last) divided by AUC(0-last).
Time Frame: as for outcome 6
Population: The pharmacokinetic (PK) population consisted of all subjects who received active investigational product, UV-4B, and had at least 1 measured concentration at a scheduled PK time after start of dosing.L/h
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h | 14.3 (15.0) | 11.4 (26.9) | 12.5 (10.1) | 13.6 (14.2) | 13.9 (12.4) | 13.7 (23.6) | 10.9 (17.6) | 11.7 (17.2)

ADVERSE EVENTS:
Time Frame: From time of the first dose administration through 9 ± 1 days after dosing
Description: Adverse events were coded by the Medical Dictionary for Regulatory Activities (MedDRA) according to system organ class (SOC) and preferred term (PT).
Arm/Group | 3 mg UV-4B | 10 mg UV-4B | 30 mg UV-4B | 90 mg UV-4B | 180 mg UV-4B | 360 mg UV-4B | 720 mg UV-4B | 1000 mg UV-4B | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 6/6 | 6/6 | 5/6 | 6/6 | 5/6 | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg UV-4B (N=6) | 10 mg UV-4B (N=6) | 30 mg UV-4B (N=6) | 90 mg UV-4B (N=6) | 180 mg UV-4B (N=6) | 360 mg UV-4B (N=6) | 720 mg UV-4B (N=6) | 1000 mg UV-4B (N=6) | Placebo (N=16)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chemical eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APTT prolonged (Investigations) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ALT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
WBC decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
WBC increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokaelemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypomagnaesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphaetemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will make the results of the study publicly available, including for purposes of national and international registration, publication, and information for medical and pharmaceutical professionals.